CLINICAL TRIAL: NCT05100550
Title: Family-based Health Education Program and Zinc Supplementation for Stunted Mother and Its Impact on Biomarker of Growth in Baby
Brief Title: Family-based Health Education Program and Zinc Supplementation for Stunted Mother
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2209210954
Record Dates: First submitted 2021-10-20; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Stunting; Maternal-Fetal Relations
Keywords: Insulin-like Growth Factor 1; Zinc; Hemoglobin; Health Education; Stunting; Low-income Family
MeSH Terms: conditions — Growth Disorders; Health Education | interventions — Zinc

STUDY DESIGN:
Intervention Model Description: One group is assigned for health education intervention and zinc supplementation, and the comparison group receives only standard antenatal care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive
  1. Health education regarding nutrition in pregnancy (including the importance of micronutrients, recognizing malnutrition, practicing breastfeeding)
  2. Screening of Low birth weight risk
  3. Zinc Supplementation 20 mg/daily from gestation week for 12 weeks, followed by 12 weeks of supplementation on the third day postpartum.
  Interventions: Dietary Supplement: Zinc
- Control (Active Comparator): Standard antenatal care for third trimester will be applied without supplementation of zinc
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Zinc — Zinc is given as written in the arm description, two hours after lunch
  Arms: Intervention
Other: Control — This group will not receive zinc
  Arms: Control

SUMMARY:
Background :

It is important to tackle the issue of malnutrition at an early stage. A stunted mother has a tendency of having adverse neonatal outcomes including growth restriction. The multidisciplinary intervention followed by micronutrient supplementation is developed to prevent these adverse outcomes. Zinc has been associated with better neonatal growth and brain growth. This study aims to assess the impact of family-based health education programs plus zinc supplementation on the important biomarker of pregnancy and neonatal growth.

Objective :

1. To assess the impact of Family-based health education programs plus zinc supplementation on the outcome of pregnancy in stunted mother
2. 1. To assess the impact of Family-based health education programs plus zinc supplementation on the outcome of neonatal growth in stunted mother

Methodology :

A Quasi-experimental study involving stunted pregnant mother with parallel intervention

Hypothesis :

Mother who receives the intervention will have the better maternal and neonatal outcome

DETAILED DESCRIPTION:
Details of Family-Based Health Education Program + Zinc :

1. Home-visit and health promotion by trained midwives
2. Supervision by health volunteer
3. Zinc Supplementation

General target population :

1. Stunted pregnant mother on the third trimester of pregnancy
2. Conducted in Primary Health Care Center

Design of Study :

two arms quasi-experimental study with one group receiving the intervention and comparison receiving standard Antenatal Care. The baseline measurement is conducted at the beginning of the third trimester, followed by the day of delivery and 6 months after delivery (for assessing the outcome of the infant). Participants are matched by certain variables

Variable :

1. Sociodemographic information
2. Food recall using Food Frequency Questionnaire

List of outcomes

1. Zinc level in breastmilk and blood of mother and infant
2. Insulin-like growth factor 1 (IGF-1) level of mother and infant
3. Hemoglobin level of mother and infant
4. Infant and placental anthropometry
5. Tumor growth Factor Beta 1 (TGF beta 1) in infant
6. Brain-derived neurotrophic factor (BDNF) in infant

Sample size using the difference between two means of neonatal birth weight who received zinc and did not receive zinc according to a study in Iran

1. Type 1 error 5%
2. Effect size: 0.4486
3. Power of study: 80%
4. With the equal allocation ratio, the total sample needed is 126

Proposed statistical analysis

1. Independent T-test
2. Linear Mixed Model

ELIGIBILITY:
Inclusion criteria

1. Body height is less than 150 cm
2. Upper Arm Circumference less than 23.5 cm
3. Family income is less than Rp 2,500,000,- following the minimum wage of targeted area
4. 24-26 weeks pregnant.

Exclusion Criteria

1. has pregnancy complications
2. multiple infants
3. refuse to follow the protocol

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study focus on a pregnant woman
Enrollment: 126 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Infant weight | changes of weight at birth up to 6 months
  This includes weight at birth, weight at 3 months and 6 months
Infant Length | changes of length at birth up to 6 months
  This includes length of body at birth, at 3 months and 6 months

SECONDARY OUTCOMES:
Hemoglobin level of mother | changes of hemoglobin level of mother from the baseline to delivery time
  Hemoglobin level of mother measured in blood using hematology analyzer
Zinc level of mother in blood | changes of Zinc in blood of mother from the baseline to 6 months after delivery
  Zinc level of mother measured in blood using hematology analyzer
Zinc level of mother in breast milk | changes of Zinc in breast milk of mother from the delivery day to 6 months after delivery
  Zinc level of mother measured in blood using atomic absorption spectrometric
Hemoglobin level of infant | changes of hemoglobin level of infant from the day of birth to 6 months
  Hemoglobin level of infant measured in blood using hematology analyzer
Insulin-like growth factor 1 (IGF-1) of mother | changes of IGF-1 level of mother from the baseline to day of delivery
  Insulin-like growth factor 1 (IGF-1) of mother measured in blood using Human IGF-1 enzyme-linked Immunosorbent Assay (ELISA)
Insulin-like growth factor 1 (IGF-1) of infant | changes of IGF-1 level of infant from the day of birth to 6 months
  Insulin-like growth factor 1 (IGF-1) of infant measured in blood using Human IGF-1 enzyme-linked Immunosorbent Assay (ELISA)
Brain-derived neurotrophic Factor (BDNF) of infant | changes of BDNF level of infant from the day of birth to 6 months
  Brain-derived neurotrophic Factor (BDNF) of infant measured in blood using enzyme-linked Immunosorbent Assay (ELISA)
Tumor Growth Factor Beta 1 (TGF beta 1) of infant | changes of TGF Beta 1 level of infant from the day of birth to 6 months
  Tumor Growth Factor Beta 1 (TGF beta 1) of infant measured in blood using enzyme-linked Immunosorbent Assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Agussalim Bukhari, MD.Ph.D, Principal Investigator — Hasanuddin University; Nurpudji A Taslim, Prof, Principal Investigator — Hasanuddin University; Aidah Baso, MD. Ph.D, Principal Investigator — Hasanuddin University; Sitti MT Chalid, MD. Ph.D, Principal Investigator — Hasanuddin University; Kadek Erika, RN, Principal Investigator — Hasanuddin University; Nasrudin Mappaware, MD, Principal Investigator — Muslim University Indonesia; Mardiana Ahmad, MD, Principal Investigator — Hasanuddin University; Firdaus Hamid, MD. Ph.D, Principal Investigator — Hasanuddin University; Suryani As'ad, Prof, Principal Investigator — Hasanuddin University; Rosdiana Natsir, Prof, Principal Investigator — Hasanuddin University; Martira Maddepungeng, MD, Principal Investigator — Hasanuddin University; Rian Pamungkas, RN, Ph.D, Principal Investigator — Esa Unggul University; Halisah Wahyuningsih, MW., Principal Investigator — Hasanuddin University; Wahyuningsih Wahyuningsih, RN, Principal Investigator — Hasanuddin University; Armiyati Nur, MW, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University Medical Research Center / HUMRC, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared accordingly

REFERENCES:
- [Background] Boskabadi H, Maamouri G, Akhondian J, Ashrafzadeh F, Boskabadi A, Faramarzi R, Heidar E, Pourbadakhshan N, Shojaei SRH, Zakerihamidi M, Vatanchi AM, Sokhtanloo M, Razaghi N, Kalani F, Ataei H, Darabi A, Mousavi MS, Hakimiakhangan S, Bagheri F. Comparison of birth weights of neonates of mothers receiving vs. not receiving zinc supplement at pregnancy. BMC Pregnancy Childbirth. 2021 Mar 6;21(1):187. doi: 10.1186/s12884-021-03598-8. PMID 33676424
- [Background] Wilson RL, Grieger JA, Bianco-Miotto T, Roberts CT. Association between Maternal Zinc Status, Dietary Zinc Intake and Pregnancy Complications: A Systematic Review. Nutrients. 2016 Oct 15;8(10):641. doi: 10.3390/nu8100641. PMID 27754451
- [Background] Prata N, Tavrow P, Upadhyay U. Women's empowerment related to pregnancy and childbirth: introduction to special issue. BMC Pregnancy Childbirth. 2017 Nov 8;17(Suppl 2):352. doi: 10.1186/s12884-017-1490-6. No abstract available. PMID 29143677
- [Background] Finch CW. Review of trace mineral requirements for preterm infants: what are the current recommendations for clinical practice? Nutr Clin Pract. 2015 Feb;30(1):44-58. doi: 10.1177/0884533614563353. Epub 2014 Dec 19. PMID 25527182
- [Background] Zahiri Sorouri Z, Sadeghi H, Pourmarzi D. The effect of zinc supplementation on pregnancy outcome: a randomized controlled trial. J Matern Fetal Neonatal Med. 2016;29(13):2194-8. doi: 10.3109/14767058.2015.1079615. Epub 2015 Sep 12. PMID 26365330